CLINICAL TRIAL: NCT00625547
Title: A Double-Blind, Randomized, Active-Controlled Multicenter Efficacy Trial for the Treatment of Patients With Restless Legs Syndrome (RLS)
Brief Title: A Study to Determine the Efficacy and Safety of Cabergoline for the Treatment of Patients With RLS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CABAS-0067-031
Record Dates: First submitted 2008-02-19; First posted 2008-02-28 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Restless Legs Syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Cabergoline; Levodopa

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: cabergoline
- 2 (Experimental)
  Interventions: Drug: levodopa

INTERVENTIONS:
Drug: cabergoline — Cabergoline oral tablets: 0.5 mg daily on Days 1 to 3, 1.0 mg daily on Days 4 to 7, 1.5 mg daily on Days 8 to 10, and 2.0 mg daily on Days 11 to 14 and then administered as a stable dose for a further 4 weeks; at Week 6, dose could be increased to 3 mg daily if patient experienced insufficient efficacy without impairing adverse events
  Arms: 1
Drug: levodopa — Levodopa oral capsules: 25 mg twice daily on Days 1 to 3, 50 mg twice daily on Days 4 to 7, 100 mg twice daily on Days 8 to 14 and then administered as a stable dose for a further 4 weeks; at Week 6, dose could be increased to 150 mg twice daily if patient experienced insufficient efficacy without impairing adverse events
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of cabergoline compared with levodopa in the treatment of patients with RLS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic RLS and had all 4 clinical manifestations of RLS
* Moderate to severe symptoms of RLS as indicated by an IRLSSG-RS total score greater than or equal to 10 and a severity at night score of greater than or equal to 4 on an 11-point RLS-6 rating scale
* No previous treatment for RLS or dissatisfaction with their current therapy

Exclusion Criteria:

* Not available

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 361 (Actual)
Dates: Start 2003-01; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the total score of the International RLS Study Group Rating Scale (IRLSSG-RS) | Week 6
Time to dropout due to a necessary change in RLS therapy because of augmentation or loss of efficacy (e.g., dose increment of study drug, switch to another therapy, or start of a drug-free period)

SECONDARY OUTCOMES:
RLS quality-of-life questionnaire | Weeks 6 and 30
Clinical Global Impression | Weeks 6 and 30
Patient Global Impression | Weeks 6 and 30
Sleep questionnaire form A | Weeks 6 and 30
IRLSSG-RS | Week 30
Safety evaluation including adverse events, clinically relevant changes in laboratory data, physical exam findings, and abnormalities observed in electrocardiogram | Weeks 2, 6, and 8 during Period 1 and every 4 weeks during Period 2
Rating of severity of RLS at night (RLS-6 scale) | Weeks 6 and 30
Rating of severity of RLS before bedtime (RLS-6 scale) | Weeks 6 and 30
Rating of severity of RLS at day when at rest and during activities, severity of daytime sleepiness (RLS-6 scales) | Weeks 6 and 30
Global rating of quality of sleep (RLS-6 scale) | Weeks 6 and 30

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- Austria (2):
  - Pfizer Investigational Site, Innsbruck
  - Pfizer Investigational Site, Vienna
- Germany (36):
  - Pfizer Investigational Site, Altötting
  - Pfizer Investigational Site, Aschaffenburg
  - Pfizer Investigational Site, Bad Honnef
  - Pfizer Investigational Site, Bad Saarow
  - Pfizer Investigational Site, Beckum
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Bochum
  - Pfizer Investigational Site, Bremerhaven
  - Pfizer Investigational Site, Dillingen
  - Pfizer Investigational Site, Duisburg
  - Pfizer Investigational Site, Düsseldorf
  - Pfizer Investigational Site, Gelsenkirchen
  - Pfizer Investigational Site, Gera
  - Pfizer Investigational Site, Göttingen
  - Pfizer Investigational Site, Halle
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Heilbronn
  - Pfizer Investigational Site, Jena
  - Pfizer Investigational Site, Kaiserslautern
  - Pfizer Investigational Site, Karlsruhe
  - Pfizer Investigational Site, Kassel
  - Pfizer Investigational Site, Köthen
  - Pfizer Investigational Site, Marburg
  - Pfizer Investigational Site, Mittweida
  - Pfizer Investigational Site, Mönchengladbach
  - Pfizer Investigational Site, Neubrandenburg
  - Pfizer Investigational Site, Oldenburg
  - Pfizer Investigational Site, Quickborn
  - Pfizer Investigational Site, Regensburg
  - Pfizer Investigational Site, Schwalmstadt
  - Pfizer Investigational Site, Schwerin
  - Pfizer Investigational Site, Stuttgart
  - Pfizer Investigational Site, Tuttlingen
  - Pfizer Investigational Site, Ulm
  - Pfizer Investigational Site, Wiesbaden
  - Pfizer Investigational Site, Wolfsburg
- Sweden (3):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Karlstad
  - Pfizer Investigational Site, Linköping
- Switzerland (3):
  - Pfizer Investigational Site, Basel, Basel
  - Pfizer Investigational Site, Bern, Canton of Bern
  - Pfizer Investigational Site, Zurich

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=CABAS-0067-031&StudyName=A%20study%20to%20determine%20the%20efficacy%20and%20safety%20of%20cabergoline%20for%20the%20treatment%20of%20patients%20with%20RLS